CLINICAL TRIAL: NCT05484011
Title: P1b, Open-Label, Safety, Tolerability, Efficacy Study of a Soluble Beta-glucan Odetiglucan in Combination w/ a CD40 Agonist (CDX-1140) in Patients w/ Metastatic Pancreatic Adenocarcinoma Whose Disease Did Not Progress During 1st-Line Chemo
Brief Title: A Maintenance Therapy Study of Odetiglucan With CDX-1140 in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: HiberCell, Inc. (Industry)
Collaborators: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PGG-PAN2111
Record Dates: First submitted 2022-07-15; First posted 2022-08-02 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — BTH1677

STUDY DESIGN:
Intervention Model Description: 3 + 3 de-escalation design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Patients will have regularly scheduled study visits on days 1, 8, and 15 of each cycle. On Day 1 patients will receive odetiglucan and CDX-1140. On Days 8 & 15 only odetiglucan. Additional study visits may be required during some cycles for safety, efficacy, and translational assessments. Patients will dose to confirmed progression, a safety event or other administrative reason requiring discontinuation; all patients are allowed to dose up to 2 years (patients continuing to derive benefit may stay on treatment longer following consultation between Investigator and Sponsor). Following discontinuation patients will be followed up to 1 year.
  Interventions: Biological: odetiglucan; Biological: CDX-1140
- Part B (Experimental): Patients will have regularly scheduled study visits on day 1 of each cycle. On Day 1 patients will receive odetiglucan and CDA-1140. Additional study visits may be required during some cycles for safety, efficacy, and translational assessments. Patients will dose to confirmed progression, a safety event or other administrative reason requiring discontinuation; all patients are allowed to dose up to 2 years (patients continuing to derive benefit may stay on treatment longer following consultation between Investigator and Sponsor). Following discontinuation patients will be followed up to 1 year.
  Interventions: Biological: odetiglucan; Biological: CDX-1140

INTERVENTIONS:
Biological: odetiglucan — Odetiglucan is a soluble, β-1,3/1,6 glucan isolated from the cell wall of a proprietary Saccharomyces cerevisiae yeast strain. Odetiglucan acts as a Pathogen-Associated Molecular Pattern (PAMP).
  Other Names: Imprime; BTH-1677; Imprime PGG
Biological: CDX-1140 — A fully human agonist anti-CD40 monoclonal antibody

SUMMARY:
The primary objective of this maintenance therapy study is to identify the maximum tolerated dose (MTD) and/ or recommended Phase 2 dose (RP2D), and evaluate the safety, tolerability, and dose-limiting toxicities (DLTs) of odetiglucan in combination with CDX-1140 in patients with metastatic PDAC with evidence of response or stable disease following a minimum of 16 and no more than 32 weeks of chemotherapy.

Up to 45 patients will be enrolled and dosed (30 patients in Part A and 15 in Part B).

DETAILED DESCRIPTION:
This is a multiple institution, open-label, 2-part Phase 1b study to determine the MTD (and/ or RP2D), safety, tolerability, and preliminary efficacy of the combination of odetiglucan and CDX-1140 for the treatment of patients with metastatic PDAC with evidence of response or stable disease during a minimum of 16 and no more than 32 weeks of therapy immediately prior to study enrollment. Part A will identify the MTD and/ or RP2D in two cohorts of patients enrolled per ABA status (Cohort 1=ABA+ and Cohort 2=ABA-) and Part B will assess an alternative dosing regimen of RP2D in an anti-beta glucan antibody ABA+, ABA- or ABA mixed population (ABA+ and ABA-) based on observations in Part A.

Product: Odetiglucan and CDX-1140 5 Protocol/Amendment No.: PGG-PAN2111, Amd.0010 Confidential - HiberCell Inc.

In Part A, a 3 + 3 de-escalation design will be used to determine the MTD of CDX-1140 when administered in combination with odetiglucan (the starting dose for CDX-1140 is that anticipated to be the recommended phase 2 dose (RP2D) based on prior Phase 1 clinical assessment). Two cohorts of patients will be enrolled (ABA+ and ABA-) and proceed independently through the 3+3 de-escalation assessment; up to 30 patients will be enrolled. The following 2 treatment cohorts will be evaluated for safety, tolerability, and preliminary efficacy:

* ABA+: Patients with ABA value ≥20 mcg/mL ABA
* ABA-: Patients with ABA value <20 mcg/mL ABA

Both cohorts will initiate at Dose Level 1 and de-escalate to Dose Level -1 based on the respective 21-day DLT period:

* Dose Level 1: Odetiglucan 4 mg/kg IV plus CDX-1140 1.5 mg/kg
* Dose Level -1: Odetiglucan 4 mg/kg IV plus CDX-1140 0.72 mg/kg Treatment will be administered in 3-week cycles. Odetiglucan will be administered weekly on Days 1, 8, and 15 of each cycle followed ~15-30 minutes later by administration of CDX-1140 1.5 mg/kg or 0.72 mg/kg IV Day 1 of each cycle.

Part B, if opened, will enroll up to 15 patients to receive odetiglucan 4 mg/kg plus the CDX-1140 RP2D identified in Part A. As in Part A, treatment will be administered in 3-week cycles, however, both odetiglucan and CDX-1140 will be administered on Day 1 of each cycle (no odetiglucan administration on Days 8 and 15 as in Part A). If the RP2D differs between Cohort 1 and Cohort 2 at the end of Part A, the Sponsor in consult with the SMC, may select a single RP2D to investigate or investigate both RP2Ds. If a larger total enrollment is required, the protocol will be amended to support.

ELIGIBILITY:
Inclusion Criteria:

1. Be age 18 years or older and has read, understood, and provided written informed consent and, if applicable, Health Insurance Portability and Accountability Act (HIPAA) authorization after the nature of the study has been fully explained and must be willing to comply with all study requirements and procedures.
2. Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma with metastatic disease.
3. Agree to be tested for peripheral blood levels of IgG anti-beta-glucan antibody (ABA) as determined by an ELISA test prior to start of study treatment.
4. Have received a minimum of 16 weeks and no more than 32 weeks of therapy (first-line chemotherapy) and experienced a CR, PR, or SD with no evidence of progression immediately before enrollment (within 14 days of first dose).

   a. Note: this requires at least durable stability or a reduction in tumor size by imaging. If a patient has demonstrated an imaging response to chemotherapy and has not progressed but had to discontinue chemotherapy prior to 16-32 weeks for a legitimate medical reason (as determined by the investigator), the patient may still be considered for the trial.
5. Have resolution of all chemotherapy-related toxicities to pre-treatment levels with exception of alopecia (which can be ongoing) and neuropathy (which can be ≤ Grade 2).
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at the time of screening.
7. Have the following laboratory values, without transfusions or growth factors, at Screening and within 14 days of the first dose of investigational agents:

   1. White blood cell count ≥2000/uL
   2. Absolute neutrophil count (ANC) ≥1.5 x 109/L.
   3. Platelet count ≥100 x 109/L.
   4. Hemoglobin ≥9 g/dL.
   5. Serum creatinine ≤1.5 mg/dL, and creatinine clearance ≥50 ml/min as measured by Cockcroft and Gault formula.
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x institution's ULN for patients with no concurrent liver metastases, OR ≤5.0 x institution's ULN for patients with concurrent liver metastases.
   7. Total bilirubin ≤1.5 x ULN, except in patients with documented Gilbert's Syndrome who must have a total bilirubin ≤3 x ULN.
   8. Serum albumin of at least 3 g/dL.
8. Have adequate coagulation function within 14 days prior to first administration of study drug on

   Day 1, as defined by either of the following criteria:
   1. International normalized ratio (INR) <1.5 × ULN OR for patients receiving warfarin or low molecular weight heparin, the patient must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these patients may exceed 1.5 × ULN if that is the goal of anticoagulant therapy
   2. Activated partial thromboplastin time (aPTT) <1.5 × ULN unless patient is receiving anticoagulant therapy, provided prothrombin time or aPTT is within therapeutic range of intended use of anticoagulants.
9. Women of childbearing potential (WOCBP) must have a negative pregnancy test (serum or urine) within the 7 days prior to study drug administration, and a negative urine pregnancy test within the 3 days before the first study drug administration, or a negative serum pregnancy test within 24 hours before the first study drug administration.
10. WOCBP and male patients who are sexually active with WOCBP must agree before receiving the first dose of study drugs to use 2 highly effective methods of contraception (including a physical barrier) during the study and for 120 days after the last dose of study drug, as described in the body of the protocol.
11. Patients must have the ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

1. Previous exposure to odetiglucan (Imprime PGG).
2. Previous exposure to CD40 antibodies or any other immunomodulatory agent for the treatment of cancer.
3. Received chemotherapy within the 14 days prior to initiation of study treatment.

   a. Concomitant antineoplastic systemic chemotherapy or biological therapy is not allowed.
4. A history of (non-infectious) pneumonitis / interstitial lung disease or has current pneumonitis / interstitial lung disease including grade 1 asymptomatic pneumonitis noted on imaging not requiring treatment.
5. Had any active or inactive autoimmune disease or syndrome (i.e., rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, inflammatory bowel disease) that required systemic treatment in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).

   a. Note: Exceptions include patients with vitiligo or resolved childhood asthma/atopy, hypothyroidism stable on hormone replacement, controlled asthma, Type I diabetes, Graves' disease, or Hashimoto's disease, or with medical monitor approval.
6. An uncontrolled concurrent illness, including an ongoing or active infection, symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina, uncontrolled hypertension, cardiac arrhythmia, interstitial lung disease or uncontrolled diabetes.
7. QT interval corrected for heart rate using Fridericia's (QTcF) method >450 msec for males and >460 msec for females.
8. A history of myocardial infarction within 6 months or a history of arterial thromboembolic event within 3 months of the first dose of investigational agent.
9. A history of human immunodeficiency virus (HIV), hepatitis B (HB), or hepatitis C, except for the following:

   1. Patients with anti-HB core antibody but with undetectable HB virus deoxyribonucleic acid (DNA) and negative for HB surface antigen
   2. Patients with resolved or treated hepatitis C virus (HCV) (i.e., HCV antibody positive but undetectable HCV RNA).
10. Received concurrent or prior use of an immunosuppressive agent within 14 days of the first dose of investigational agent, with the following exceptions and notes:

    1. Systemic steroids at physiologic doses (equivalent to dose of 10 mg oral prednisone) are permitted.
    2. Intranasal, inhaled, topical intra-articular, and ocular corticosteroids with minimal systemic absorption are permitted.
    3. Transient course of steroids may be approved by the Medical Monitor on a case by case basis, dependent on dose, timing and reason.
11. Active, untreated central nervous system (CNS) metastases or a history of clinically manifested central nervous system (CNS) metastases.

    a. Note: Patients with brain metastases identified at Screening may be rescreened after the lesion(s) have been appropriately treated; patients with treated brain metastases should be neurologically stable for 4 weeks post-treatment and prior to study enrollment, and off corticosteroids for at least 2 weeks before administration of study drugs, and treated lesions should demonstrate no new growth on the re-screening scan
12. Known or suspected leptomeningeal disease or cord compression. Product: Odetiglucan and CDX-1140 11 Protocol/Amendment No.: PGG-PAN2111, Amd.000 Confidential - HiberCell Inc.
13. Had major surgery as determined by the investigator within 4 weeks before the first dose of study drug. Surgery requiring local/epidural anesthesia must be completed at least 72 hours before study drug administration and patients should be recovered.
14. Other prior malignancy, except for adequately treated basal or squamous cell skin cancer or in situ cancers; or any other cancer from which the patient has been disease-free for at least 3 years.
15. Received another investigational agent within the shorter of 4 weeks or 5 half-lives before the first dose of investigational agents.
16. Received a live attenuated vaccine within 28 days before the first dose of investigational agent, and patients, if enrolled, should not receive live vaccines during the study or for 30 days after the last dose of investigational agent.
17. Females who are pregnant or lactating or who intend to become pregnant during participation in the study are not eligible to participate.
18. Known alcohol or drug abuse.
19. Any clinically significant psychiatric, social, or medical condition that, in the opinion of the investigator, could increase the patient's risk, interfere with protocol adherence, or affect the patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Within 24 months of last patient enrolled
  Determination of MTD of odetiglucan + CDX-1140

SECONDARY OUTCOMES:
Duration of Response | Within 24 months of last patient enrolled
  Duration of response following treatment with odetiglucan + CDX-1140
Overall Response Rate | Within 24 months of last patient
  ORR per RECIST v1.1 and immune-RECIST (iRECIST) following treatment with odetiglucan + CDX-1140
Median Progression Free Survival and Progression Free Survival at 6 Months | Within 36 months of last patient enrolled
  Median progression free survival and progression free survival at 6 months by RECIST v1.1 following treatment with odetiglucan + CDX-1140
Median Overall Survival and Overall Survival at 1 Year | Within 36 months of last patient enrolled
  Median OS and OS at 1 year following treatment with odetiglucan + CDX-1140

CONTACTS AND LOCATIONS:
Overall Officials: Mark O'Hara, Study Chair — University of Pennsylvania
Locations (4):
- United States (4):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No